CLINICAL TRIAL: NCT02229409
Title: Effectiveness of the Walking Intervention Walkadoo: A Randomized Controlled Pilot Trial in an Employee Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MeYou Health, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WD-PILOT-2014
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Observation only, no behavioral intervention
- Intervention (Experimental): Intervention Walkadoo.
  Interventions: Behavioral: Walkadoo

INTERVENTIONS:
Behavioral: Walkadoo — Walkadoo is a MeYou Health, LLC product.
  Arms: Intervention

SUMMARY:
This study evaluates the product Walkadoo to determine whether it effectively increases walking behavior in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older;
* Healthways employees based in Franklin, TN with an email account with the company;
* Provide informed consent and complete eligibility questionnaires

Exclusion Criteria:

* Current or prior use of the intervention Walkadoo
* Presence of a chronic condition that affects walking
* Projected inability to access the internet for 4 consecutive days or longer during the study
* Non-adherence to device wear during baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Average steps per day | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nathan K Cobb, MD, Study Director — Georgetown University
Locations (1):
- MeYou Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poirier J, Bennett WL, Jerome GJ, Shah NG, Lazo M, Yeh HC, Clark JM, Cobb NK. Effectiveness of an Activity Tracker- and Internet-Based Adaptive Walking Program for Adults: A Randomized Controlled Trial. J Med Internet Res. 2016 Feb 9;18(2):e34. doi: 10.2196/jmir.5295. PMID 26860434